CLINICAL TRIAL: NCT00105859
Title: Preventing Pressure Ulcers in Veterans With Spinal Cord Injury (SCI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Garber, Susan - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 01-151
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2005-06

CONDITIONS: Spinal Cord Injury; Pressure Ulcers
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer | interventions — Educational Status; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: Education and Counseling

INTERVENTIONS:
Behavioral: Education and Counseling

SUMMARY:
Pressure ulcers are a serious, costly, and life-long complication of spinal cord injury (SCI). Pressure ulcer prevalence has been estimated at between 17 and 33% among persons with SCI residing in the community. Epidemiological studies have found that 36-50% of all persons with SCI who develop pressure ulcers will develop a recurrence within the first year after initial healing (Carlson et al., 1992; Fuhrer et al., 1993; Goldstein, 1998; Niazi et al., 1997; Salzberg et al. 1998). Recurrence rates have ranged from 21% to 79%, regardless of treatment (Schryvers et al., 2000; Goodman et al., 1999; Niazi et al., 1997). Pressure ulcer treatment is expensive. Surgical costs associated with pressure ulcer treatment can exceed $70,000 per case (Braun et al., 1992). VA administrative (National Patient Care Database, NPCD) data indicate that 41% of inpatient days in the SCI population are accounted for by either primary or secondary diagnoses of pressure ulcers or 23% of SCI inpatient days if restricted to primary diagnoses of pressure ulcers. Pressure ulcer recurrence has been associated with many factors including previous pressure ulcer surgery (Niazi et al., 1997). Although little data exist describing the factors associated with recurrence following surgery, some investigators reported recurrence rates of 11%-29% in cases with post-operative complications and 6% to 61% in cases without post-operative complications (Mandrekas & Mastorakos, 1992; Relander & Palmer, 1988; Disa et al., 1992). In a retrospective study of 48 veterans with SCI, investigators reported a 79% recurrence rate following surgery (Goodman et al., 1999).

DETAILED DESCRIPTION:
Background:

Pressure ulcers are a serious, costly, and life-long complication of spinal cord injury (SCI). Pressure ulcer prevalence has been estimated at between 17 and 33% among persons with SCI residing in the community. Epidemiological studies have found that 36-50% of all persons with SCI who develop pressure ulcers will develop a recurrence within the first year after initial healing (Carlson et al., 1992; Fuhrer et al., 1993; Goldstein, 1998; Niazi et al., 1997; Salzberg et al. 1998). Recurrence rates have ranged from 21% to 79%, regardless of treatment (Schryvers et al., 2000; Goodman et al., 1999; Niazi et al., 1997). Pressure ulcer treatment is expensive. Surgical costs associated with pressure ulcer treatment can exceed $70,000 per case (Braun et al., 1992). VA administrative (National Patient Care Database, NPCD) data indicate that 41% of inpatient days in the SCI population are accounted for by either primary or secondary diagnoses of pressure ulcers or 23% of SCI inpatient days if restricted to primary diagnoses of pressure ulcers. Pressure ulcer recurrence has been associated with many factors including previous pressure ulcer surgery (Niazi et al., 1997). Although little data exist describing the factors associated with recurrence following surgery, some investigators reported recurrence rates of 11%-29% in cases with post-operative complications and 6% to 61% in cases without post-operative complications (Mandrekas & Mastorakos, 1992; Relander & Palmer, 1988; Disa et al., 1992). In a retrospective study of 48 veterans with SCI, investigators reported a 79% recurrence rate following surgery (Goodman et al., 1999).

Objectives:

The purpose of this project was to identify effective interventions for reducing recurrent pressure ulcers, a severe costly complication in veterans with SCI. The effect of an educational and structured telephone counseling follow-up program on prevention and health care utilization were being evaluated. Hypotheses included the following: 1) After discharge from the hospital for treatment of a severe healed pelvic pressure ulcer, patients receiving the education and structured telephone counseling intervention would be significantly less likely to develop a new or recurrent severe (e.g., Stage III or IV), pelvic (defined for this study as occurring in the sacrum, coccyx, trochanter, or ischium) pressure ulcer than those receiving customary care. 2) Admissions and inpatient days for severe pelvic pressure ulcers will be significantly lower for veterans receiving the education and structured telephone counseling intervention when compared to those receiving customary care.

Methods:

Veterans admitted to 6 VA SCI Centers for medical and/or surgical treatment of a Stage III or IV pelvic pressure ulcer (sacrum, coccyx, trochanter or ischium) were randomly assigned to (1) an Intervention Group consisting of education plus structured telephone counseling follow-up or (2) a Customary Care (Control) group. Intervention Group subjects received a cognitive behavioral intervention based on the Trans-theoretical Stages of Change Model, which is designed to help individuals identify ways of improving health behaviors. On admission, interviewers collected information on demographics, health status/well being, locus of control, pressure ulcer knowledge, readiness-to-change, and health beliefs/practices. Some of these measures were re-administered prior to randomization and at 9 and 18 months post-discharge. Health care utilization was monitored for all participants for the length of the study. The primary outcome (dependent) variables were (1) the occurrence or non-occurrence of another pelvic pressure ulcer within 18 months of discharge following healing and, (2) for individuals who develop pressure ulcers during the study period, time to recurrence. Intervention Group participants were expected to have fewer pressure ulcer-related admissions and, if admitted, a shorter hospital stay. Secondary outcomes included health care utilization, pressure ulcer prevention knowledge, medical and psychological health status, health beliefs and practices, and quality of life. Multi-variate logistic models are being used to examine factors associated with recurrence and to evaluate the impact of recurrence on health care utilization.

Status:

A total of 64 patients were randomized in this study, 33 to customary care and 31 to the intervention group. Most were male, white, married and had their SCI at the thoracic level resulting in paraplegia. Mean time to recurrence was 114.50 days for the total randomized subjects. All data from all 15 questionnaires are being analyzed and will be put into a manuscript for publication at a future time.

ELIGIBILITY:
Inclusion Criteria:

SCI more than 1 year duration, admitted to VA for treatment of a stage III or IV pressure ulcer, access to telephone for follow-up, understands english, cognitively intact

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Garber, MA BS, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (6):
- United States (6):
  - VA Medical Center, Augusta, Augusta, Georgia
  - Memphis, TN, Memphis, Tennessee
  - Houston VA Medical Center, Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Clement J. Zablocki VAMC, Milwaukee, Wisconsin

REFERENCES:
- [Result] Guihan M, Garber SL, Bombardier CH, Durazo-Arizu R, Goldstein B, Holmes SA. Lessons learned while conducting research on prevention of pressure ulcers in veterans with spinal cord injury. Arch Phys Med Rehabil. 2007 Jul;88(7):858-61. doi: 10.1016/j.apmr.2007.03.014. PMID 17601465
- [Result] Guihan M, Garber SL, Bombardier CH, Goldstein B, Holmes SA, Cao L. Predictors of pressure ulcer recurrence in veterans with spinal cord injury. J Spinal Cord Med. 2008;31(5):551-9. doi: 10.1080/10790268.2008.11754570. PMID 19086713
- [Derived] Guihan M, Bombardier CH. Potentially modifiable risk factors among veterans with spinal cord injury hospitalized for severe pressure ulcers: a descriptive study. J Spinal Cord Med. 2012 Jul;35(4):240-50. doi: 10.1179/2045772312Y.0000000016. PMID 22925750